CLINICAL TRIAL: NCT04477733
Title: Effect of Butorphanol on Colonoscopy for Patients With Postoperative Visceral Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: wj20200710
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Colonoscopy
Keywords: Butorphanol, Visceral pain, Propofol, Gastroscopy, Colonoscopy
MeSH Terms: conditions — Visceral Pain | interventions — Butorphanol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butorphanol group (Experimental)
  Interventions: Drug: Butorphanol Injection
- control group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Butorphanol Injection — Inject 10 μg/kg of butorphanol, then propofol is injected until the patient's eyelash reflex disappears before performing colonoscopy
  Arms: Butorphanol group
Drug: Saline — Inject saline and propofol until the patient's eyelash reflex disappears before performing colonoscopy
  Arms: control group

SUMMARY:
The total incidence of abdominal pain after colonoscopy is almost 50%. Butorphanol is a mixed opioid receptor agonist-antagonist, which has strong sedative and analgesic effects. This clinical study aims to explore the effectiveness and safety of butorphanol combined with propofol for colonoscopy to reduce postoperative visceral pain, and provide a basis for improving the quality of surgery and comfortable medical treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-11
* patients performing colonoscopy
* sign the informed consent

Exclusion Criteria:

* BMI>30, pregnant
* diabetes
* depression
* patients dependent on opioids
* hypertension poorly controlled
* serious complications of important organs
* obvious abdominal pain before colonoscopy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
visceral pain | 10 minutes after recovery
  VAS score of visceral pain

SECONDARY OUTCOMES:
visceral pain at 20 and 30 minutes after recovery | 20 and 30 minutes after recovery
  VAS score of visceral pain

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

REFERENCES:
- [Derived] Wang J, Wang X, Liu H, Han R. Effect of butorphanol on visceral pain in patients undergoing gastrointestinal endoscopy: a randomized controlled trial. BMC Anesthesiol. 2023 Mar 28;23(1):93. doi: 10.1186/s12871-023-02053-9. PMID 36977981